CLINICAL TRIAL: NCT01252836
Title: Randomized, Prospective, Pilot Study Evaluating a Temporary Skin Substitute (AWBAT-D) Versus the Standard of Care in the Postoperative Treatment of Split-thickness Skin Graft Donor Sites
Brief Title: Study Evaluating AWBAT-D Versus the Standard of Care of Split-thickness Skin Graft Donor Sites
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: P.I decided to prematurely end this study.
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Director of Center for Wound Healing, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-160
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Healing of Donor Site; Pain Level

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Treatment with Tegaderm
  Interventions: Device: AWBAT-D
- AWBAT-D (Experimental): Application of AWBAT-D on donor site.
  Interventions: Device: AWBAT-D

INTERVENTIONS:
Device: AWBAT-D — Application of AWBAT-D bioengineered device

SUMMARY:
Use of AWBAT-D on split thickness skin graft sites will reduce healing time and pain level.

DETAILED DESCRIPTION:
The study is designed as a randomized-controlled trial to examine split thickness skin graft donor wound site healing using AWBAT-D compared to current standard of care: Tegaderm. This will involve randomizing subjects to treatment with the AWBAT-D dressing or Tegaderm and monitoring outcomes. The AWBAT-D device has collagen and we hypothesize that the wounds treated with it will heal faster and with a decreased pain level. The purpose of this study is to evaluate if there are differences in outcomes between AWBAT-D and Tegaderm in healing split thickness skin graft donor sites.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subjects requiring a split-thickness skin graft with a wound size between 5 and 50cm2 and a depth between 12-18um.
3. Ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study.

Exclusion Criteria:

1. Subjects < 18 years of age
2. Subjects with an allergy to porcine products.
3. Subjects undergoing STSG with a wound size less than 5 cm2 or greater than 50cm2.
4. Subjects undergoing STSG with a wound depth of less than 12um or greater than 18um.
5. Subjects undergoing repeat skin graft harvesting at the same donor site.
6. Has active malignant disease of any kind. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
7. Subjects participating in any other trials involving the split-thickness skin graft donor site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time for donor site to heal with AWBAT-D | 6 weeks
  As compared to current standard of care, Tegaderm.

SECONDARY OUTCOMES:
Pain at donor site | 6 weeks
  Pain at donor site is less than that of standard of care treatment, Tegaderm.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Attinger, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital Center for Wound Healing, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data was not collected for use in future research and will not be shared.